CLINICAL TRIAL: NCT03116945
Title: 68Gallium Citrate Imaging in Newly Diagnosed Hepatocellular Carcinoma
Brief Title: Novel Gallium Imaging in Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Nasrin Ghesani, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20150001631
Record Dates: First submitted 2016-04-28; First posted 2017-04-17 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: PET/CT; 68Gallium Citrate; Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Drug; 68Gallium Citrate (Experimental): Procedure: PET/CT Imaging
  Interventions: Drug: 68Gallium Citrate

INTERVENTIONS:
Drug: 68Gallium Citrate — Procedure: PET/CT Imaging
  Other Names: Scintigraphy

SUMMARY:
The aim of the present study is to validate the uptake of novel, positron emitting radiotracer, 68Gallium Citrate in hepatocellular carcinoma(HCC). The investigators also aim to evaluate the sensitivity of 68Gallium (68Ga)-citrate positron emission tomography/computed tomography (PET/CT) for the identification of intrahepatic HCC lesions in comparison with existing modalities: computed tomography (CT) alone and magnetic resonance imaging (MRI). The investigators expect that 68Ga-citrate PET/CT will offer a sensitive functional imaging modality for identification of HCC lesions in the liver. The investigators intend to use the results of this preliminary study to fuel further studies in the utility of 68Ga-citrate PET/CT for HCC treatment monitoring.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a malignancy of the liver with very high mortality. Management of HCC often involves interventional and surgical therapies that distort surrounding liver morphology. For this reason, current morphologic imaging techniques following these therapies often fail to distinguish between residual tumor and post-therapeutic morphologic changes. Therefore, there is the need for an effective imaging technique in therapy monitoring for HCC.

Functional imaging techniques are commonly used in other cancers for effective therapy monitoring. Functional imaging in HCC with single photon emitting gallium radioisotopes has been explored in the past but have not been used routinely due to poor resolution of images. 68Gallium-citrate PET/CT can generate high resolution images that specifically target HCC cells regardless of liver morphology. This makes 68Gallium-citrate PET/CT an ideal imaging modality for HCC following therapies that distort liver morphology.

Before determining its efficacy in therapy monitoring, The investigators aim to demonstrate the ability for 68Gallium-citrate PET/CT to localize known intrahepatic HCC lesions.

In this pilot study, 18 subjects with newly diagnosed HCC will be recruited. Each subject will undergo a 68Gallium-citrate PET/CT scan within 6 weeks of radiographic diagnosis. Foci of abnormal radiotracer uptake on these scans will be tabulated and compared to clinically-indicated morphologic imaging. The investigators expect that 68Gallium-citrate PET/CT will offer a sensitive functional imaging modality for identification of HCC lesions in the liver. The investigators intend to use the results of this preliminary study to form the basis for grant applications to extra-mural funding agencies. These subsequent grant applications will focus on further studies in the utility of 68Gallium-citrate PET/CT for HCC therapy monitoring and metastatic work-up.

ELIGIBILITY:
Inclusion Criteria:

* At least one biopsy-confirmed or Liver Imaging Reporting and Data System (LI-RADS)- 5 HCC lesion, diagnosed within the past 6 weeks.
* Lesion size greater than or equal to 3cm
* At least one triple-phase CT or MRI of the liver prior to medical or surgical therapy

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Current somatic or psychiatric disease/condition that may interfere with the objectives and assessments of the study.
* Inability to consent
* Prior medical or surgical therapy for HCC, including chemoembolization, radiofrequency ablation, and lobectomy
* Known or suspected hypersensitivity to metals or gallium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2016-06 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Uptake of positron emitting radiotracer, 68Gallium Citrate will be measured in the lesions of hepatocellular carcinoma. | One Year
  For each subject, presence and location of abnormal radiotracer localization will be recorded. Tumor volume will be measured on CT, MRI, and PET/CT images using the MIM software. Region-of-interest (ROI) will be drawn around each area of morphologic abnormality on PET/CT images to calculate a mean standardized uptake value (SUV), a maximum SUV, and a target-to-background ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Nasrin Ghesani, MD, Principal Investigator — Rutgers University
Locations (1):
- Rutgers New Jersey Medical School, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Gharib AM, Thomasson D, Li KC. Molecular imaging of hepatocellular carcinoma. Gastroenterology. 2004 Nov;127(5 Suppl 1):S153-8. doi: 10.1053/j.gastro.2004.09.029. PMID 15508079